CLINICAL TRIAL: NCT04960657
Title: The Hemodynamic Effects of PACAP38 After Glibenclamide Administration in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Lili Kokoti, MD, PhD student, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H19065735
Record Dates: First submitted 2021-05-24; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Migraine; Headache; Pain
Keywords: Glyburide; Physiological Effects of Drugs; Hypoglycemic Agents
MeSH Terms: conditions — Migraine Disorders; Headache; Pain | interventions — Glyburide; Pituitary Adenylate Cyclase-Activating Polypeptide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, cross-over, placebo-controlled design in healthy volunteers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACAP38 and glibenclamide (Active Comparator): Participants will receive glibenclamide after PACAP38 infusion
  Interventions: Drug: glibenclamide; Drug: PACAP38
- PACAP38 and placebo (Active Comparator): Participants will receive placebo after PACAP38 infusion
  Interventions: Drug: glibenclamide; Drug: PACAP38

INTERVENTIONS:
Drug: glibenclamide — Oral administration of glibenclamide/placebo. To investigate the role of PACAP38 on cranial arteries in healthy volunteers after glibenclamide/placebo administration .
Drug: PACAP38 — PACAP38 infusion
  Other Names: Pituitary adenylate cyclase activating polypeptide-38

SUMMARY:
To investigate the hemodynamic effects of PACAP38 after glibenclamide administration.

DETAILED DESCRIPTION:
22 healthy participants will randomly be allocated to receive PACAP38 infusion followed by glibenclamide or placebo on two different days.

The aim of the study is to investigate the vascular effect of PACAP38 after glibenclamide administration.

Repeated measurements covering the arteria radialis (RA), superficial temporal artery (STA) and middle cerebral artery (MCA) before and after PACAP38 infusion and glibenclamide/placebo administration

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes.
* 18-60 years.
* 50-100 kg.
* Women of childbearing age must use adequate contraception

Exclusion Criteria:

* A history of serious somatic or psychiatric disease
* Migraine or any other type of headache (except episodic tension-type headache less than 5 days per month)
* Daily intake of any medication except contraceptives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Headache | Time of headache measurements is from before (-20 minutes) and up to 12 hours after PACAP38 infusion
  Headache intensity will be recorded by numerical rating scale (NRS) from 0 to 10 (0, no headache; 1, a feeling of pressure; 10, worst imaginable headache).

SECONDARY OUTCOMES:
Changes in the arterial radialis (RA), superficial temporal artery (STA) and middle cerebral artery (MCA). | Time of measurements is baseline and repeatedly every 20 minutes for 260 minutes.
  Repeated measurements covering the diameter of RA, STA and MCA before and after PACAP38 infusion and glibenclamide/placebo administration measured by centimeter (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No